CLINICAL TRIAL: NCT04486573
Title: Identification of Early Cardiac Injury From Radiation Therapy Using Cardiac Magnetic Resonance Imaging
Brief Title: Cardiac Effects From Radiation Therapy by MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-0537.cc; NCI-2020-06349 (Other: CTRP)
Record Dates: First submitted 2020-07-10; First posted 2020-07-24 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Radiation Treatment; Cancer; Cardiotoxicity
MeSH Terms: conditions — Neoplasms; Cardiotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CMRI (Other): Clinical data will be collected regarding cardiac risk factors, cancer type, and cancer treatment.
  CMRI will be performed:
  * Within 2 weeks before the first fraction of radiation therapy (RT)
  * Within 1 week of the final fraction of RT (before or after)
  Any patient with a pre-RT and post-RT MRI scan will be considered evaluable.
  Pre- and post-RT CMRI parameters will be compared.
  3D reconstructed CMR images will be co-registered with RT treatment plans to assess for spatial associations.
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance Imaging — A cardiac MRI is a painless imaging test that uses radiowaves, magnets, and a computer to create detailed pictures of the heart.

SUMMARY:
The investigators will identify 10 patients in the department of radiation oncology who will receive standard of-care radiation therapy, and the treating radiation oncologist anticipates a mean left ventricular dose of at least 5 Gy. Patients will be evaluated by CMRI before and within one week of the completion of RT. We will compare the pre- and post-RT CMRI scans to identify changes related to radiation exposure. Our primary endpoint will be changes in myocardial strain. Secondary endpoints will include other CMRI parameters.

DETAILED DESCRIPTION:
Cardiac toxicity is a significant cause of morbidity and mortality in cancer survivors after radiation therapy (RT) to the chest. Typically, cardiotoxicity is identified years after radiation exposure. Emerging clinical data show that subclinical injury can be identified immediately after treatment. Early identification of subclinical injury may enable intervention to reduce the risk of progression to clinically significant toxicity. The investigators hypothesize that cardiac magnetic resonance imaging (CMRI) will detect early cardiac injury after RT and that imaging changes will be associated regionally with cardiac radiation dose.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. 18 - 100 years of age
4. KPS ≥ 70 or ECOG ≥ 1
5. Will receive RT using computed tomography (CT)-based treatment planning that will involve delivery of dose to the heart
6. Estimated by the treating radiation oncologist at the time of simulation to have a mean left ventricular dose of at least 5 Gy

Exclusion Criteria:

1. Previous history of RT to the thorax or breast
2. Implanted device that is non-MRI compatible or any implanted device in chest
3. Known gadolinium contrast allergy or other contraindication to CMRI scan. Patients needing sedation or medication for claustrophobia or anxiety will not be excluded from participating.
4. Found to be pregnant or breast-feeding
5. Known history of atrial fibrillation or frequent ventricular or atrial premature beats
6. Known history of chronic kidney disease (such as, but not limited, to a glomerular filtration rate < 60mL/min)
7. History of coronary artery disease or myocardial disease
8. History of hypertension, requiring >1 antihypertensive agent to maintain blood pressure <140/90
9. Known history of valvular stenosis or regurgitation of > moderate severity
10. Known history of heart failure (defined as baseline New York Heart Association Class III or IV (see Appendix A)
11. Systolic blood pressure < 90mmGy
12. Pulse < 50/minute
13. Known history of pulmonary hypertension or elevated right ventricular systolic pressures.
14. Suspicion or diagnosis of amyloidosis
15. Suspicion or diagnosis of hemochromatosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Change in myocardial strain | 2 years
  Assess for a change in myocardial strain, as measured by CMRI scans performed before and after RT

SECONDARY OUTCOMES:
T1 pre- and post-contrast values | 2 years
  Measured by scans performed before and after RT
Extracellular volume fraction | 2 years
  Measured by scans performed before and after RT
T2 values | 2 years
  Measured by scans performed before and after RT
Late gadolinium enhancement | 2 years
  Measured by scans performed before and after RT
Left ventricular ejection fraction | 2 years
  Measured by scans performed before and after RT
End diastolic volume | 2 years
  Measured by scans performed before and after RT
End systolic volume | 2 years
  Measured by scans performed before and after RT
Left atrial volume | 2 years
  Measured by scans performed before and after RT
Wall thickness | 2 years
  Measured by scans performed before and after RT
Left ventricular mass index | 2 years
  Measured by scans performed before and after RT

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Milgrom, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No